CLINICAL TRIAL: NCT04764799
Title: HEAVEN Criteria: a Monocentric Prospective Observational Study to Validate the Prediction of Difficult Airway for In-Hospital Emergency Airway Management
Brief Title: HEAVEN Criteria: Prediction of Difficult Airway for In- Hospital Emergency Airway Management
Status: Completed | Type: Observational
Sponsor: Thomas Riva (Other)
Responsible Party: Sponsor-Investigator, Thomas Riva, Prof. Dr. med., Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: HEAVEN_BRN; 2020-02458 (Registry Identifier: swissethics)
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Failure
Keywords: Emergency Medicine; Intubation, Intratracheal; Anesthesiology; Rapid Sequence Induction; Difficult Airway; Prediction Tool
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Rapid Sequence Induction and Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients that need emergency rapid sequence inductions: Patients of all ages who need emergency rapid sequence inductions due to their medical condition performed by the staff of the Department of Anaesthesiology and Pain Medicine at the Bern University Hospital.
  We defined "emergency" as a non scheduled intervention with immediate (or maximum up to 6 hours after announcement) need of general anaesthesia (e.g. trauma patients with need for emergency surgery) and therefore appropriate fastening is not possible.
  Interventions: Procedure: Rapid sequence induction
- Patients that need scheduled rapid sequence inductions: Patients of all ages who need scheduled rapid sequence inductions due to their medical condition performed by the staff of the Department of Anaesthesiology and Pain Medicine at the Bern University Hospital.
  Patients of this cohort have a scheduled intervention and therefore can fasten meals for at least 6 hours before induction of general anaesthesia.
  Interventions: Procedure: Rapid sequence induction

INTERVENTIONS:
Procedure: Rapid sequence induction — Rapid sequence induction starts with the administration of rapid acting intravenous narcotics, opioids and neuromuscular blockage and avoids whenever possible positive-pressure ventilation after induction of anesthesia.

SUMMARY:
The HEAVEN criteria were found valid to predict difficult airways during preclinical emergency intubations in a retrospective study. The acronym stands for Hypoxemia, Extremes of size, Anatomic abnormalities, Vomit/blood/fluid, Exsanguination/anaemia, and Neck mobility issues. This is a monocentric prospective observational study to assess the validity of the HEAVEN criteria in the in-hospital setting at a level I adult and pediatric emergency university-based hospital.

DETAILED DESCRIPTION:
Emergency intubations are prone to present a difficult airway. A difficult airway can lead to prolonged intubation time and to hypoxemia in situations where oxygenation is not possible that can finally result in hypoxic cardiac arrest and irreversible brain damage caused by hypoxic ischemic encephalopathy.

Tools to predict difficult airways are rather poor concerning specificity and sensitivity. A score to predict difficult airway developed in the pre-clinical setting are the HEAVEN criteria. The acronym HEAVEN stands for: Hypoxemia, Extremes of size, Anatomic abnormalities, Vomit/blood/fluid, Exsanguination/anaemia, and Neck mobility issues and does not need patients' cooperation. It has been recently validated in the pre-clinical emergency setting and was found to be useful.

The study aim is to evaluate if the HEAVEN criteria are suitable to be used to predict difficult airway in in-hospital emergency intubation to finally increase patients' safety during rapid sequence induction (RSI).

This prospective observational single-centre study in emergency intubation will consecutively recruit all patients of all ages who need RSI due to their medical condition performed by the staff of the Department of Anaesthesiology and Pain Medicine at the Bern University Hospital. We will record data that are gathered during routine patient care and stored primarily in the departmental anaesthesia information systems.

The primary objective is to validate if the HEAVEN criteria, an existing prehospital difficult airway prediction tool, is able to predict airways difficulties during RSI in the clinical in-hospital setting. The secondary objective is, to assess the subcomponent of the HEAVEN criteria and if differences and adaptations are needed comparing it to the prehospital setting.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients of all ages who need an in-hospital rapid sequence intubation (RSI) performed by the staff of the Department of Anesthesiology and Pain Medicine
* Given general consent or delayed obtained general consent after the procedure
* English, German or French speaking patients

Exclusion Criteria:

• Patients without informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who need rapid sequence intubation due to their medical condition at the Bern University Hospital are screened if they fulfill the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 2800 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Patients with first-attempt success rate of RSI | 1 hour
  Every attempt starts with the insertion of a laryngoscope blade over the lips and ends with a blocked tube in the trachea and measuring of carbon dioxide (CO2)
Patients with difficulty of intubation | 1 hour
  Rated on a scale by the airway manager: easy, difficult, not possible

SECONDARY OUTCOMES:
Overall success rate of rapid sequence induction (RSI) | 1 hour
  All RSI during the study period are analyzed for success (If intubation is possible or not)
Patients with first-attempt success without desaturation SpO2 <92% during RSI | 1 hour
  Saturation will be measured and recorded during the whole intervention and analyzed for the time of the RSI.
Total attempts of intubation in a patient | 1 hour
  Every attempt starts with the insertion of a laryngoscope blade over the lips and ends with a blocked tube in the trachea and measuring of CO2
Cormack & Lehane grade (C&L) or Percentage of Glottis Opening (POGO) in a patient | 1 hour
  C&L for direct laryngoscopy or POGO for video laryngoscopy will be recorded for every intubation
Lowest and highest recorded value of patients' heart rate (HR) during RSI | 1 hour
  Heart rate will be measured and recorded during the whole intervention and analyzed for the time of the RSI.
Lowest and highest recorded value of patients' blood-pressure (BP) during RSI | 1 hour
  BP will be measured and recorded during the whole intervention and analyzed for the time of the RSI.
Lowest and highest recorded value of patients' oxygen saturation (SpO2) during RSI | 1 hour
  SpO2 will be measured and recorded during the whole intervention and analyzed for the time of the RSI.
Patients with use of vasoconstrictors during RSI | 1 hour
  Use of vasoconstrictors will be recorded during the whole intervention and analyzed for the time of the RSI.
Patients with use of devices/ techniques for intubation | 1 hour
  Use of:
  * supraglottic airway device (SAD)
  * intubation guides (Frova, S-Guide)
  * video laryngoscopy (VL) or direct laryngoscopy, shape and size of the blade, flexible scope
  * rigid stylets ("C-MAC VS", "Bonfils")
  * intubation over SAD
  * emergency front of neck access (eFONA)
Patients with use and type of neuromuscular blockage agent | 1 hour
  Yes / No, if Yes, specify: Succinylcholine, Rocuronium, Atracurium, other
Patient's demographics | 1 hour
  Patient's age, gender, weight and size
Type of planned procedure | 1 day
  type of surgery by discipline (e.g. ear, nose and throat (ENT), visceral, orthopedic, heart, urology, gynecology) and specification (e.g. appendectomy)
Place of intubation | 1 day
  The place where the intubation is performed. Either operation room (OR) or outside OR
Time of intubation | 1 hour
  the exact time (HH:MM:SS) in central european time of the induction of the RSI
Level of airway manager | 1 hour
  nurse, resident or attending anaesthesiologist
Endotracheal tube (ETT) | 1 hour
  Type and size of the used ETT(s) during the RSI attempt(s)
Patients with airway-related injuries like blood, damage to tissue, lips or teeth caused directly during intubation | 1 hour
  Will be directly recorded if occurred during the RSI by the airway manager or team
Patients with airway-related complains like hoarseness or problems with swallowing until 24 hours after intubation reported subjectively by the patient | 1 day
  All patients will be visited in the first 24 hours after anaesthesia if they report subjectively airway-related complains like hoarseness or problems with swallowing until 24 hours after intubation and evaluated by an anaesthesiologist or further referred to an ENT specialist
Patients with suspicion of aspiration during RSI | 1 day
  Newly recorded suspicion of aspiration during intubation will be recorded by the airway team

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD, Prof., Study Chair — Department of Anaesthesiology and Pain Medicine, Inselspital, Bern University Hospital, Switzerland
Locations (1):
- University Hospital Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No